CLINICAL TRIAL: NCT05364515
Title: Randomized Clinical Trial, Controlled to Conventional Treatment, to Evaluate the Efficacy of Plasma Rich in Growth Factors (PRGF) for the Treatment of Lichen Sclerosus Atrophicus of the Vulva
Brief Title: Plasma Rich in Growth Factors (PRGF) for the Treatment of Lichen Sclerosus Atrophicus of the Vulva
Acronym: PRGF
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The PI left the participating center and, due to the care load of the service to which she belonged, no clinician was able to take charge of the clinical trial. The clinical trial was never started, no participating subjects were included.
Sponsor: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTIIMD-01-EC/217LIQUEN
Record Dates: First submitted 2022-04-12; First posted 2022-05-06 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Lichen Sclerosus of Vulva
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional treatment (Active Comparator): 0.05% Clobetasol propionate
  Interventions: Drug: Clobetasol Propionate
- PRGF (Experimental): 0.05% Clobetasol propionate + PRGF
  PRGF: 4 infiltrations (first two months) + topical administration (from third month)
  Interventions: Drug: PRGF; Drug: Clobetasol Propionate

INTERVENTIONS:
Drug: PRGF — Plasma Rich in Growth Factors (PRGF) is a mixture of proteins and growth factors obtained from the blood of the patient.
  Four PRGF infiltrations (two weeks between each infiltration). Then, application of topical PRGF serum (on alternate basis)
  Arms: PRGF
Drug: Clobetasol Propionate — 0.05 propionate clobetasol: daily (first month), alternate (second moth), twice per week (from third month)

SUMMARY:
Lichen sclerosus is a chronic dermatosis of the skin and semimucous membranes, characterized by the presence of well-defined atrophic white papules or plaques, which appear mainly on the skin of the anogenital region of both sexes, and less frequently on the skin of the trunk. , mainly affecting postmenopausal women. There is no absolutely effective treatment. Only potent topical corticosteroids control symptoms and improve outcomes, although prolonged use can increase skin atrophy. In severe vulvar lesions, 0.05% clobetasol propionate is indicated, followed by a less potent topical corticosteroid. Relapses often occur if treatment is discontinued altogether, but respond well to reintroduction of treatment.

Plasma Rich in Growth Factors (PRGF®) is a mixture of autologous proteins, prepared from a certain volume of platelet-rich plasma obtained from a small volume of blood, which does not contain leukocytes. To date, there have been no studies evaluating PRGF® treatment in vulvar lichen sclerosus. However, there are several publications that assess the efficacy of PRPs as a treatment for vulvar lichen sclerosus. This clinical study has been designed with the aim of evaluating the efficacy of PRGF® in reducing the main symptoms of vaginal lichen sclerosus atrophicus.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Woman with symptoms associated with LEA confirmed by histological study
* Being 1 month without prior treatment in the affected area as a washing period
* Availability of observation during the treatment period
* Signature of the informed consent

Exclusion Criteria:

* Acute somatic disease
* Infection in the intervention area or active systemic infection
* History of cancerous or precancerous lesions in the intervention area
* In active treatment with other local treatments in the intervention area
* Under active treatment with immunosuppressants and/or anticoagulants
* History of allergies to blood derivatives
* Previous diagnosis of coagulopathies
* Regular and continuous treatment with NSAIDs
* Positive markers for HCV, AfHBs, HIV-I/II or PT
* Pregnancy or women of childbearing age not taking contraceptive measures
* Lactating women
* Treatment with monoclonal antibodies
* Liver failure
* Any inability to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Evolution of quality of life measured by Skindex-29 index | 6 months
  Quality of life in patients with cutaneous disease (Skindex-29 index). Values from 0 to 116. Lower scores mean a better outcome
Evolution of quality of life measured by Skindex-29 index | 8 months
  Quality of life in patients with cutaneous disease (Skindex-29 index). Values from 0 to 116. Lower scores mean a better outcome

SECONDARY OUTCOMES:
Evolution of quality of life measured by Skindex-29 index | 1 and 3 months
  Quality of life in patients with cutaneous disease (Skindex-29 index). Values from 0 to 116. Lower scores mean a better outcome
Evolution of response to treatment at 1, 3, 6 and 8 months through the clinical scale of vulvar lichen sclerosus (CSS) | 1, 3, 6 and 8 months
  Values: from 0 to 40. Lower scores mean a better outcome.
Evolution of pain at 1, 3, 6 and 8 months measured through the visual analog pain scale (VAS) | 1, 3, 6 and 8 months
  Values: from 0 to 40. Lower scores mean a better outcome.
Evolution of the improvement at 1, 3, 6 and 8 months through the patient's global impression (PGI-I) | 1, 3, 6 and 8 months
  Evolution of the improvement at 1, 3, 6 and 8 months through the patient's global impression (PGI-I)
Evolution of clinical improvement at 1, 3, 6 and 8 months through the investigator's global assessment (IGA) | 1, 3, 6 and 8 months
  Evolution of clinical improvement at 1, 3, 6 and 8 months through the investigator's global assessment (IGA)
Frequency of recurrences at 6 and 8 months of treatment | 6 and 8 months
  Frequency of recurrences at 6 and 8 months of treatment
Frequency of complications | 1, 3, 6 and 8 months
  Frequency of complications
Platelet concentration | 0 months
  Platelet concentration measurement in whole blood and PRGF fraction
Platelet recovery | 0 months
  Platelet enrichment (PRGF vs. whole blood)
Presence of leukocyte | 0 months
  % of leukocyte in PRGF fraction

IPD SHARING:
Plan to Share IPD: No